CLINICAL TRIAL: NCT07071532
Title: A Phase 1 Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of ABBV-932 in Healthy Adult Subjects
Brief Title: A Study to Assess Adverse Events and How Oral ABBV-932 Moves Through the Body When Given With Oral Itraconazole in Healthy Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M24-966
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-932; Itraconazole
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-932 with Itraconazole (Experimental): Participants will receive ABBV-932 in Period 1 followed by Itraconalzole in combination with ABBV-932 in Period 2.
  Interventions: Drug: ABBV-932; Drug: Itraconazole

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule
Drug: Itraconazole — Oral Capsule
  Other Names: ITZ

SUMMARY:
This study will assess the adverse events and how oral ABBV-932 moves through the body when given with oral Itraconazole in healthy Adults participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* History: of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of suicidal ideation within one year prior to study treatment administration and/or history of suicidal behavior or non-suicidal self-injury within two years prior to study treatment administration as evidenced by any "yes" answer to questions on the Columbia - Suicide Severity Rating Scale (C-SSRS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  Cmax of ABBV-932 and active metabolites DCAR and DDCAR
Time to Cmax (Tmax) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  Tmax of ABBV-932 and active metabolites DCAR and DDCAR
Observed plasma concentration at the end of a dosing interval (Ctrough) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  Ctrough of ABBV-932 and active metabolites DCAR and DDCAR
Apparent terminal phase elimination rate constant (β) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  (β) of ABBV-932 and active metabolites DCAR and DDCAR
Terminal Phase Elimination Half-Life (t1/2) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  Terminal phase elimination half-life of ABBV-932 and active metabolites DCAR and DDCAR
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  AUCt of ABBV-932 and active metabolites DCAR and DDCAR
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-932 and active metabolites DCAR and DDCAR | Up to approximately 29 days
  AUCinf of ABBV-932 and active metabolites DCAR and DDCAR
Number of Participants Experiencing Adverse Events | Up to approximately 61 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 276951, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-966